CLINICAL TRIAL: NCT03995407
Title: 100% Whey Protein Based Diet In Enhancing Pressure Ulcer Healing- A Pilot Randomized Controlled Trial.
Brief Title: 100% Whey Protein Based Diet In Enhancing Pressure Ulcer Healing.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resourcing issues impacted by COVID-19 pandemic.
Sponsor: St Luke's Hospital, Singapore (Other)
Responsible Party: Principal Investigator, JIANG SONG'EN, JEFFREY, Principal Investigator, St Luke's Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-03-2019-01-03
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Pressure Ulcer
Keywords: Pressure ulcer; Whey protein; Wound healing
MeSH Terms: conditions — Pressure Ulcer | interventions — Peptamen

STUDY DESIGN:
Intervention Model Description: Parallel 2-arm pilot randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants in the control arm will receive "usual care".
  Interventions: Other: Usual Care
- 100% Whey Protein (Experimental): Participants will receive 100% Whey Protein oral nutritional supplements.
  Interventions: Dietary Supplement: Peptamen®

INTERVENTIONS:
Dietary Supplement: Peptamen® — Participants in the intervention arm will be categorised into those who are not currently taking oral nutritional supplement and those who are currently on oral nutritional supplements. Those who are not currently taking oral nutritional supplement will be started on Peptamen® while those who are currently on oral nutritional supplements will have to convert to Peptamen® solely. The dietician will determine the amount of Peptamen® required per day based on the recommendations of the product information. Should the participant's daily protein requirement not be met be Peptamen® alone, the dietician will recommend additional whey protein to be added in the form of Beneprotein® Instant Protein Powder. Beneprotein® is a concentrated source of high-quality whey protein that can be added to most foods, liquids or enteral formulas.
  Arms: 100% Whey Protein
Other: Usual Care — Participants receive "usual care". They will be categorised into those who are not currently taking oral nutritional supplement and those who are currently on oral nutritional supplements (non-100% whey i.e. not on Peptamen® or Beneprotein®). They will consume their regular diet in accordance with the dietician's recommendations.
  Arms: Control

SUMMARY:
This study seeks to evaluate if a 100% whey protein based diet enhances pressure ulcer healing.

DETAILED DESCRIPTION:
A pressure ulcer is defined as an area of localized damage to the skin and underlying tissues caused by pressure, shear, friction, and/or a combination of these. The most common sites for pressure ulcers are the sacrum, heels, ischial tuberosities, greater trochanters, and lateral malleoli.

In Singapore, the prevalence of pressure ulcers was 18.1%, while the incidence was 8.1% in a tertiary hospital in Singapore in 2002. With a rapidly ageing population in Singapore, the prevalence of pressure ulcers is expected to increase further.

Pressure ulcers are associated with serious medical complications, prolonged hospital stay and frequent re-admissions. Patients with pressure ulcers generally have significantly poorer physical function, are less able to perform self-care, and are less mobile. A new pressure ulcer is estimated to increase a patient's hospital stay by nearly a factor of five. Furthermore, pressure ulcers are also correlated with more than two fold rates of increased mortality independent of the source of the ulcer. Pressure ulcers are one of the patient safety indicators reflecting quality of life according to the Agency for Healthcare Research and Quality. Besides affecting the quality of life of patients, pressure ulcers are also associated with the increased utilisation of healthcare resources resulting in a high cost burden to healthcare systems worldwide.

Pressure ulcers occur in individuals with limited mobility due to pressure, or pressure in combination with shear, which decreases circulation and causes tissue damage. Elderly patients and patients with specific predisposing conditions such as hip fractures are particularly at risk. In addition, patients whom are malnourished are not only at risk of pressure ulcers but also have impaired wound healing. Patients with pressure ulcers tend to have negative energy balance and current guidelines recommend the assessment of nutritional status when progress for pressure ulcers closure does not occur and the use of oral nutritional supplements when an oral diet is not sufficient to meet requirements. In particular, nutritional care in wound healing should be directed at ensuring adequate supply of proteins and calories. Major guidelines currently recommend a minimum calorie intake of 30-35 kilocalories per kg per day and protein intake of 1.25-1.5g per kg per day for adults with a pressure ulcer who are assessed as being at risk of malnutrition.

Currently, there is paucity of studies demonstrating the effect whey protein has on wound healing in humans. The effect of whey protein on wound healing has only been studied in diabetic rats which has shown to accelerate closure and the healing process of their wounds. It was postulated that the healing property of whey was due to its ability to limit prolonged inflammation (reduction in IL-6, TNF-alpha, IL-1b and IL-10) and elevating the antioxidant defence system (by up-regulating glutathione and superoxide dismutase).

Whey protein comprises of 20% of the protein content in cow's milk as compared to casein which makes up the remainder of 80%. Whey is made up of immunoglobulins, lactoalbumins, lactoferrin, cysteine and other minor proteins. Compared to casein, whey has rapid gut clearance as it is readily absorbed, has higher nutritional value, maintains and increases lean body mass and has shown to have greater muscle protein accrual in the elderly. Moreover, whey has positive immuno-modulatory effects and is able to maintain better glycaemic control in diabetics due to its lower post-prandial glycaemia, greater stimulation of incretin production and direct insulinotropic effect.

At present, Peptamen® is the only product available in Singapore that contains 100% hydrolysed whey protein. It is a commercially available peptide-based diet (classified under "medical foods" by the US Food and Drug Administration) that provides complete nutrition. It is hypoallergenic (lactose- and gluten-free), appropriate for those with gastrointestinal maldigestion and/or malabsorption and can be used for total nutrition support via oral or tube feeding. We hypothesize that a 100% whey protein based diet (Peptamen®) enhances pressure ulcer healing.

ELIGIBILITY:
Inclusion Criteria:

1. Any age, gender or ethnicity.
2. Admitted for subacute wound care.
3. Diagnosed with stage 3 or 4 pressure ulcer.
4. Wound surface area > 4cm2.

Exclusion Criteria:

1. Prognosis of less than 1 year.
2. Diagnosed with osteomyelitis of the wound.
3. Allergy to soy or corn.
4. Chronic Kidney Disease Stage 4 or 5.
5. Participants who are already consuming oral nutritional supplements and are not willing to convert to Peptamen® if allocated to the intervention arm.
6. Participants who are currently consuming Peptamen® or another 100% whey protein oral nutritional supplement.
7. Dislikes the taste of milk.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Percentage Reduction in Wound Surface Area | 4 weeks
  Percentage reduction in wound surface area = [Surface area at baseline - Surface area after 4 weeks] / [Surface area at baseline] %
Pressure Ulcer Score for Healing (PUSH) Score | 4 weeks
  The Pressure Ulcer Scale for Healing (PUSH Tool) was developed by the National Pressure Ulcer Advisory Panel (NPUAP) as a quick, reliable tool to monitor the change in pressure ulcer status over time. The total score ranges from 0 (best condition) to 17 (worst condition) and is derived from 3 parameters (product of length and width of wound, exudate amount, and tissue type).

SECONDARY OUTCOMES:
Amount of Peptamen® and Beneprotein® consumed | 4 weeks
  Measured in grams.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jiang Song'en, MBBS, Principal Investigator — St. Luke's Hospital
Locations (1):
- St Luke's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No